CLINICAL TRIAL: NCT02247193
Title: Botulinum Toxin to Improve Cosmesis of Primary Cleft Lip Repair
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Matthew Greives, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSC-MS-14-0335
Record Dates: First submitted 2014-09-17; First posted 2014-09-23 (Estimated); Results first posted 2021-11-03 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Cleft Lip; Scarring; Cleft Palate
Keywords: Botulinum Toxin; Botox; Craniofacial deformity
MeSH Terms: conditions — Cleft Lip; Cicatrix; Cleft Palate | interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Botulinum Toxin (Experimental): Injection of botulinum toxin into cleft lip at time of surgical repair.
  Interventions: Drug: Botulinum Toxin Type A
- Saline (Placebo Comparator): Injection of normal saline into cleft lip at time of surgical repair.
  Interventions: Drug: Normal Saline Injection

INTERVENTIONS:
Drug: Botulinum Toxin Type A — Injection of botulinum toxin at the time of surgery at cleft lip repair site. Botulinum toxin will be injected intraoperatively at 4 standardized sites in the cleft lip during surgical repair.
  Arms: Botulinum Toxin
Drug: Normal Saline Injection — Injection of normal saline into cleft lip at time of surgical repair. Saline will be injected intraoperatively at 4 standardized sites in the cleft lip during surgical repair.
  Arms: Saline

SUMMARY:
Objective: To determine if the use of botulinum toxin during primary cleft lip repair improves the cosmetic appearance of the cleft lip scar

ELIGIBILITY:
Inclusion Criteria:

* complete unilateral cleft lip with or without cleft palate
* planned for a primary cleft lip repair

Exclusion Criteria:

-bilateral cleft lip

Max Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2020-01-13 (Actual); Study Completion 2020-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaecel O Shah, MD, Principal Investigator — UTHealth
Locations (1):
- Memorial Hermann Hospital, Houston, Texas, United States

REFERENCES:
- [Background] Pascual-Pascual SI, Pascual-Castroviejo I. Safety of botulinum toxin type A in children younger than 2 years. Eur J Paediatr Neurol. 2009 Nov;13(6):511-5. doi: 10.1016/j.ejpn.2008.10.006. Epub 2008 Nov 25. PMID 19036619
- [Background] Galarraga IM. Use of botulinum toxin in cheiloplasty: A new method to decrease tension. Can J Plast Surg. 2009 Fall;17(3):e1-2. doi: 10.1177/229255030901700313. PMID 20808741
- [Background] Alvarez CM, De Vera MA, Chhina H, Williams L, Durlacher K, Kaga S. The use of botulinum type A toxin in the treatment of idiopathic clubfoot: 5-year follow-up. J Pediatr Orthop. 2009 Sep;29(6):570-5. doi: 10.1097/BPO.0b013e3181b2b3d4. PMID 19700985
- [Background] Gassner HG, Sherris DA, Friedman O. Botulinum toxin-induced immobilization of lower facial wounds. Arch Facial Plast Surg. 2009 Mar-Apr;11(2):140-2. doi: 10.1001/archfacial.2009.3. No abstract available. PMID 19289689
- [Background] Christiansen G, Mohney BG, Baratz KH, Bradley EA. Botulinum toxin for the treatment of congenital entropion. Am J Ophthalmol. 2004 Jul;138(1):153-5. doi: 10.1016/j.ajo.2004.02.023. PMID 15234303
- [Background] Sherris DA, Gassner HG. Botulinum toxin to minimize facial scarring. Facial Plast Surg. 2002 Feb;18(1):35-9. doi: 10.1055/s-2002-19825. PMID 11823931
- [Background] Sykes JM. Management of the cleft lip deformity. Facial Plast Surg Clin North Am. 2001 Feb;9(1):37-50. PMID 11465005
- [Background] Seibert RW. Bilateral cleft nasal repair. Facial Plast Surg. 2000;16(1):69-78. doi: 10.1055/s-2000-7328. PMID 11802349
- [Background] Millard DR Jr. Embryonic rationale for the primary correction of classical congenital clefts of the lip and palate. Ann R Coll Surg Engl. 1994 May;76(3):150-60. PMID 8017808
- [Background] Witt PD, Hardesty RA. Rotation-advancement repair of the unilateral cleft lip. One center's perspective. Clin Plast Surg. 1993 Oct;20(4):633-45. PMID 8275629
- [Background] Lee JS, Lee KB, Lee YR, Choi YN, Park CW, Park SD, Jung DH, Lee CS. Botulinum Toxin Treatment on Upper Limb Function in School Age Children With Bilateral Spastic Cerebral Palsy: One Year Follow-up. Ann Rehabil Med. 2013 Jun;37(3):328-35. doi: 10.5535/arm.2013.37.3.328. Epub 2013 Jun 30. PMID 23869330

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Botulinum Toxin | Saline
Started | 15 | 15
Number Who Underwent Cleft Lip Repair Surgery | 15 | 15
Number Who Received Botox or Placebo | 15 | 15
Number Who Completed the 6-month Follow up | 15 | 15
Number Who Completed the 12-month Follow up | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Botulinum Toxin | Saline | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: days] | 129.53 (27.27) | 135.67 (17.41) | 132.6 (22.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 14
  Male | 6 | 10 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 1 | 2
  Caucasian | 8 | 6 | 14
  Hispanic | 6 | 8 | 14
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 15 | 30
Number of Participants with Syndromic Cleft Lip [Count of Participants; unit: Participants] | 1 | 0 | 1
Number of Participants with Presurgical Nasoalveolar Molding (PNAM) [Count of Participants; unit: Participants] | 10 | 12 | 22
Number of Participants with Complete Cleft Lip [Count of Participants; unit: Participants] | 13 | 13 | 26
Number of Participants with Unilateral Cleft Lip [Count of Participants; unit: Participants] | 14 | 15 | 29
Number of Participants with Cleft Palate [Count of Participants; unit: Participants] | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Hypertrophic Scarring (HTS) as Assessed by Score on the Manchester Scar Scale (MSS) Rated by Blinded Plastic Surgeons
Description: The Manchester Scar Scale (MSS) assesses color match to surrounding skin, skin texture, contour, and distortion, and total MSS score ranges from 4 to 14, with a higher score indicating worse scarring. Scars were analyzed by three blinded plastic surgeons, who evaluated frontal and basal photographs of participants. The median of the three surgeon scores per participant was first calculated, and then the median all medians was calculated per arm.
Time Frame: 6 months
Population: Only 9 in the Botulinum Toxin arm and 11 in the Saline arm were analyzed for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Botulinum Toxin | Saline
Number analyzed (Participants) | 9 | 11
score on a scale | 7 [7 to 10] | 9 [8 to 10]

2. Primary Outcome: Hypertrophic Scarring (HTS) as Assessed by Score on the Manchester Scar Scale (MSS) Rated by Blinded Plastic Surgeons
Description: as for outcome 1
Time Frame: 12 months
Population: Only 9 in the Botulinum Toxin arm and 11 in the Saline arm were analyzed for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Botulinum Toxin | Saline
Number analyzed (Participants) | 9 | 11
score on a scale | 7 [6.5 to 7] | 9 [6.5 to 9.5]

3. Primary Outcome: Hypertrophic Scarring (HTS) as Assessed by Score on the Modified Scar Rating Scale (MSRS) Rated by Blinded Plastic Surgeons
Description: The Modified Scar Rating Scale (MSRS) assesses surface appearance, scar height, and color mismatch, and total MSRS score ranges from 3 to 12, with a higher score indicating worse scarring. Scars were analyzed by three blinded plastic surgeons, who evaluated frontal and basal photographs of participants. The median of the three surgeon scores per participant was first calculated, and then the median all medians was calculated per arm.
Time Frame: 6 months
Population: Only 9 in the Botulinum Toxin arm and 11 in the Saline arm were analyzed for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Botulinum Toxin | Saline
Number analyzed (Participants) | 9 | 11
score on a scale | 7 [6.0 to 8.0] | 8 [6.0 to 8.0]

4. Primary Outcome: Hypertrophic Scarring (HTS) as Assessed by Score on the Modified Scar Rating Scale (MSRS) Rated by Blinded Plastic Surgeons
Description: as for outcome 3
Time Frame: 12 months
Population: Only 9 in the Botulinum Toxin arm and 11 in the Saline arm were analyzed for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Botulinum Toxin | Saline
Number analyzed (Participants) | 9 | 11
score on a scale | 6 [6.0 to 7.0] | 7 [6.5 to 7.5]

5. Primary Outcome: Hypertrophic Scarring (HTS) as Assessed by Score on the Manchester Scar Scale (MSS) Rated by Crowdsourced Raters
Description: The Manchester Scar Scale (MSS) assesses color match to surrounding skin, skin texture, contour, and distortion, and total MSS score ranges from 4 to 14, with a higher score indicating worse scarring. Scars were analyzed by crowdsourced raters via Amazon Mechanical Turk. The crowdsourced raters evaluated frontal and basal photographs of participants. 100 unique responses were elicited per participant. The mean of all crowdsourced ratings for each arm is reported per arm.
Time Frame: 6 months
Population: Only 9 in the Botulinum Toxin arm and 11 in the Saline arm were analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Botulinum Toxin | Saline
Number analyzed (Participants) | 9 | 11
score on a scale | 7.40 (0.74) | 8.29 (0.47)

6. Primary Outcome: Hypertrophic Scarring (HTS) as Assessed by Score on the Manchester Scar Scale (MSS) Rated by Crowdsourced Raters
Description: as for outcome 5
Time Frame: 12 months
Population: Only 8 in the Botulinum Toxin arm and 12 in the Saline arm were analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Botulinum Toxin | Saline
Number analyzed (Participants) | 8 | 12
score on a scale | 7.48 (0.78) | 7.72 (0.64)

7. Primary Outcome: Hypertrophic Scarring (HTS) as Assessed by Score on the Modified Scar Rating Scale (MSRS) Rated by Crowdsourced Raters
Description: The Modified Scar Rating Scale (MSRS) assesses surface appearance, scar height, and color mismatch, and total MSRS score ranges from 3 to 12, with a higher score indicating worse scarring. Scars were analyzed by crowdsourced raters via Amazon Mechanical Turk. The crowdsourced raters evaluated frontal and basal photographs of participants. 100 unique responses were elicited per participant. The mean of all crowdsourced ratings for each arm is reported per arm.
Time Frame: 6 months
Population: Only 9 in the Botulinum Toxin arm and 11 in the Saline arm were analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Botulinum Toxin | Saline
Number analyzed (Participants) | 9 | 11
score on a scale | 5.96 (0.74) | 6.74 (0.5)

8. Primary Outcome: Hypertrophic Scarring (HTS) as Assessed by Score on the Modified Scar Rating Scale (MSRS) Rated by Crowdsourced Raters
Description: as for outcome 7
Time Frame: 12 months
Population: Only 8 in the Botulinum Toxin arm and 12 in the Saline arm were analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Botulinum Toxin | Saline
Number analyzed (Participants) | 8 | 12
score on a scale | 6.01 (0.75) | 6.19 (0.69)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Botulinum Toxin | Saline
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

LIMITATIONS AND CAVEATS:
Small sample size; inconsistency in acquiring post-op photos for some; 12 month analysis may be skewed by Botox's short duration of action; crowdsourced raters were not a generalized sample of the population

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-02-17): https://cdn.clinicaltrials.gov/large-docs/93/NCT02247193/Prot_SAP_000.pdf